CLINICAL TRIAL: NCT03448653
Title: Contribution of Narrow Band Imaging (NBI) for the Characterization of Scalloped Polyps
Brief Title: Contribution of Narrow Band Imaging (NBI) for the Characterization of Scalloped Polyps (NBI POLYPES COLIQUES)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment, advances in technology
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHD010-17
Record Dates: First submitted 2018-02-21; First posted 2018-02-28 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Polyps of Colon
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy; Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colonoscopy with NBI (Experimental)
  Interventions: Other: Colonoscopy with NBI

INTERVENTIONS:
Other: Colonoscopy with NBI — Colonoscopy with NBI

SUMMARY:
This prospective bicentric trial aims to evaluate the diagnostic performance of the characterization of scalloped polyps less than 20 millimeter in NBI (Narrow Band Imaging) in patients with screening colonoscopy.

The NBI is a so-called "virtual" electronic staining technique available on conventional OLYMPUS endoscopes without additional intervention.

The colonoscopy procedure for each patient will not be different from a conventional colonoscopy examination with excision of all polyps visualized and anatomopathological analysis, except for a short time of analysis in NBI for each polyp detected before excision to classify the polyp in existing endoscopic classifications (ie NICE classification for adenomatous polyps and WASP classification for festooned polyps).

ELIGIBILITY:
Pre-inclusion criteria:

* Major patient with a colonoscopy scheduled in one of the participating hospitals (CHD Vendée and CHU Nantes).
* Patient who agreed to participate in the study and gave his express consent
* Patient affiliated with a social security system or beneficiary of a scheme

Inclusion Criteria:

* Patient with 1 or more polyps less than 20 mm observed during colonoscopy

Exclusion Criteria:

* Patient with an emergency colonoscopy for ongoing digestive bleeding or occlusion symptoms
* Patient with chronic inflammatory bowel disease (IBD): Crohn's disease or unclassified colitis
* Patient with familial adenomatous polyposis
* Pregnant or lactating woman
* Minor patient
* Major patient under tutorship, curatorship, or deprived of liberty
* Patient unable to understand protocol and / or give express consent
* Patient not affiliated with a social security system or beneficiary of such a scheme
* Patient hospitalized or treated without their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent MACE, Study Director — Centre Hospitalier Départemental Vendée
Locations (2):
- France (2):
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier Universitaire Nantes, Nantes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Colonoscopy With NBI
Started | 314
Completed | 314
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colonoscopy With NBI
Number analyzed (Participants) | 312
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Not regulatory
  Not Hispanic or Latino | NA — Not regulatory
  Unknown or Not Reported | 312
Region of Enrollment [Number; unit: participants]
  France | 312

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the NBI Compared to the Anatomopathological Analysis (= Reference Method)
Description: Number of polyps characterized as scalloped (NICE II-) by NBI relative to the number of polyps characterized as scalloped in standard histology
Time Frame: An average of 1 month
Population: All polyps with histological analysis available in eligible patients
Measure: Number (95% Confidence Interval); unit: proportion of positive cases
Units Other Than Participants: polyps
Arm/Group | Colonoscopy With NBI
Number analyzed (Participants) | 312
Number analyzed (polyps) | 522
proportion of positive cases | 0.844 [0.803 to 0.879]

ADVERSE EVENTS:
Description: Death, serious adverse event and other (not serious adverse event) were not assessed for the study
Arm/Group | Colonoscopy With NBI
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT03448653/Prot_SAP_000.pdf